CLINICAL TRIAL: NCT04292717
Title: Precision Medicine in the Rehabilitation of Locomotor Function: Individual Gait Profiles for Deficit-specific Training Strategies in Spinal Disorders
Brief Title: Deficit-specific Training in Spinal Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-00247
Record Dates: First submitted 2020-02-20; First posted 2020-03-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries; Multiple Sclerosis; Gait Disorders, Neurologic; Training; Neurorehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Multiple Sclerosis; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deficit-oriented training group (Active Comparator)
  Interventions: Behavioral: Gait training
- Non-specific, standardised walking training group (Active Comparator)
  Interventions: Behavioral: Gait training

INTERVENTIONS:
Behavioral: Gait training — All participants will receive training three times a week for 6 weeks (18 training sessions) at the University Hospital Balgrist, Spinal Cord Injury Centre. Each exercise session will last for 1 hour and will be conducted and supervised by an experienced physical therapist.

SUMMARY:
Impairments of walking function after spinal cord lesion due to, for example, inflammation, ischemia or trauma are exceptionally diverse. Depending on the size, location and completeness of the spinal cord lesion, gait dysfunction is often multifactorial, arising from weakness of leg muscles, sensory impairments or spasticity. Locomotor function in humans with spinal cord damage can be improved through training. However, there are no evidence-based guidelines for the treatment of gait dysfunctions and no excepted standards of gait training in this large and heterogeneous group of patients. A lack of evidence-based guidance and standardisation prevents the development of optimal training programs for patients with spinal cord damage and rather broad and subjective clinical judgement is applied to determine patient care. Objective and quantitative techniques like three-dimensional (3D) full-body movement analysis capable of identifying the most relevant determinants of gait dysfunction at the single-patient-level are not yet implemented as diagnostic tool to guide physical therapy in this heterogeneous group of patients. The objective of this project is to further advance current clinical locomotor training strategies by applying a deficit-oriented gait training approach based on subject-specific, objective gait profiles gleaned from 3D gait analysis in chronic, mildly to moderately gait-impaired individuals with spinal cord damage due to inflammation (in multiple sclerosis, MS) or with traumatic or ischemic spinal cord injury (SCI; motor incomplete). Within a parallel-group clinical trial, gait impaired subjects will be characterized by detailed kinematic 3D gait analysis and either trained according to their individual deficits or treated with non-specific, standard walking therapy for six weeks. It is hypothesized that individually adapted, deficit-oriented training is superior in improving walking function than purely task-related, ambulatory training in patients with spinal cord damage. This project may pave the way to more efficient training approaches in subjects with spinal cord damage by transferring and implementing modern gait assessment techniques into clinical neurorehabilitation and to move towards individual, patient-tailored locomotor training programs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Diagnosis of chronic spinal cord injury (>6 months cervical or thoracic motor incomplete traumatic or non-traumatic (AIS C, D) above T12 or diagnosis of either primary- progressive, secondary-progressive, or relapsing-remitting multiple sclerosis as defined by the revised McDonald criteria for at least 3 months and with at least one spinal cord lesion as verified in clinical MRI images
* Able to walk without assistance or devices on the treadmill and 10m over ground, but must have impaired walking function as demonstrated by neurological examination.

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Current orthopaedic problems of lower limbs
* History of major cardiac condition (e.g., infarction, insufficiency (NYHA II-IV))
* History of major pulmonary condition (e.g., chronic obstructive pulmonary disease GOLD II-IV)
* Current major depression or psychosis
* MS exacerbation within 3 months prior to the screening or at any time during the screening period
* Participation in another training study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
Six minute walk test (6MWT) | Change from screening at 10 weeks

SECONDARY OUTCOMES:
MS-patients: Expanded disability status scale (EDSS) | Change from screening at 10 weeks
  neurological score, range from 0 to 10, lower values better than higher values
SCI-patients: ISNCSCI by the American Spinal Injury Association (ASIA protocol) | Change from screening at 10 weeks
  Perceptions of light touch (LT) and pinprick (PP) stimuli are scored as 0 for absent, 1 for impaired and 2 for normal (range for sum score for pin prick and light touch: 0-112). Motor function is scored on the Medical Research Council Scale of 0 for total paralysis to 5 for normal strength. Ten muscles are tested bilaterally and individual muscle scores are added together, yielding an ASIA motor score that ranges from 0 to 100. For all assessments higher scores are better than lower scores.
SCI-patients: Walking index for Spinal Cord Injury (WISCI II) | Change from screening at 10 weeks
  Range from 0-20, higher values are better than lower values.
MS-/ SCI-patients: Six-minute walk test (6MWT) | 10 weeks
MS-patients. Timed 25-foot walk (T25FW) | Change from screening at 10 weeks
SCI-patients: Timed 10-meter walk test (10MWT) | Change from screening at 10 weeks
MS-/ SCI-patients: Timed up and go test (TUG) | Change from screening at 10 weeks
MS-/ SCI-patients: Kinematic measures on treadmill | Change from screening at 6 and 10 weeks
  A set of key kinematic parameters will be quantified describing leg, trunk and arm movements during walking on a treadmill including range of motion (in degrees) of hip, knee and ankle joints.
MS-/ SCI-patients: Kinetic measures | Change from screening at 6 and 10 weeks
  A set of key kinetic parameters will be quantified describing forces of weight loading for both feet using pedobarography.
MS-/ SCI-patients: Electromyographic measures | Change from screening at 6 and 10 weeks
  EMG measures include timing of leg muscle activity during walking on treadmill.
MS-/ SCI-patients: 12-item WS for walking function (questionnaire) | Change from baseline at 10 weeks
  Questionnaire, range from 12-60 points, lower values are better than higher values.
MS-/ SCI-patients: Time to swim 10m | Change from baseline at 6 weeks
MS-/ SCI-patients: Kinematic parameters of leg movements during swimming (activity sensors) | Change from baseline at 6 weeks
  A set of key kinematic parameters will be quantified describing leg movements during swimming including range of motion (in degrees) of hip, knee and ankle joints.
MS-/SCI-patients: Spinal Cord Independence Measure (SCIM-III) | Change from screening at 10 weeks
MS-/ SCI-patients: Magnetic resonance imaging (MRI) | Change from baseline at 10 weeks
MS-/ SCI-patients: Magnetic resonance spectroscopy (MRS) | Change from baseline at 10 weeks
MS-/ SCI-patients: over ground gait kinematics during clinical walking tests (activity sensors) | Change from baseline at 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik Balgrist, Zurich, Switzerland